CLINICAL TRIAL: NCT00410787
Title: Safety and Tolerability of Long-Term Administration of Dilaudid SR (Hydromorphone HCI) in Cancer Pain
Brief Title: Safety and Tolerability of Long-term Administration of OROS Hydromorphone HCI (Slow Release) in Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013264
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Analgesics, Opioid; Pain
Keywords: Chronic cancer pain; OROS hydromorphone HCI (slow release); long-term repeated dosing
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: OROS hydromorphone HCI (slow release)

SUMMARY:
The primary purpose of this study was to characterize the pain control achieved with long-term repeated dosing of OROS hydromorphone (slow release) in patients with chronic cancer pain and the secondary purpose was to characterize the effects of pain on the patients' quality of life with long-term, repeated dosing of OROS hydromorphone (slow release) taken by patients with chronic cancer pain.

DETAILED DESCRIPTION:
Study DO-118X was a phase-3, multicenter, open-label extension study in adult patients with cancer pain who had successfully completed Study DO-118 with dose-stable pain control taking at least 8 mg of OROS hydromorphone (slow release) or its equivalent morphine sulfate SR (slow release) dosage. Patients were started on the dose of OROS hydromorphone equivalent to the opioid dose on which they had achieved dose-stable pain control in the SR (slow release) phase of Study DO-118. Patients returned to their study clinic once a month for 1 year. Dosage adjustments to study medications and breakthrough pain medication were permitted. OROS hydromorphone HCI (slow release) tablets in 8, 16, 32 and 64mg doses administered orally every 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic cancer pain, and who have successfully completed the OROS hydromorphone SR (slow release) study, DO-118
* Patients must have been in dose-stable pain control in the last two days of the slow release phase of the study
* Patients who require at least 8mg of OROS hydromorphone slow release every 24 hours for the management of chronic cancer pain

Exclusion Criteria:

* Pain which is not considered to be potentially responsive to opioids
* Gastrointestinal disease of sufficient severity to be likely to interfere with oral analgesia including: dysphagia, vomiting, no bowel movement or bowel obstruction due to impaction within the 5 days prior to the start of the trial, severe gut narrowing that may affect the absorption or transit of orally administered drugs, particularly the insoluble OROS outer coating
* Any patient in whom the risks of treatment with hydromorphone outweigh the potential benefits. Such risk categories include: raised intracranial pressure, hypotension, hypothyroidism, asthma, reduced respiratory reserve, prostatic hypertrophy, hepatic impairment, renal impairment, elderly and debilitated, convulsive disorders and Addison's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Study results indicated that long-term treatment with OROS hydromorphone can be useful in the management of persistent, moderate-to-severe chronic pain in patients with cancer

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA